CLINICAL TRIAL: NCT07011979
Title: SNU IBD Cohort Study : Searching for Characterization of High Risk Populations for Developing Inflammatory Bowel Disease (SNU PREVENT)
Brief Title: SNU IBD Cohort Study : Searching for Characterization of High Risk Populations for Developing Inflammatory Bowel Disease
Acronym: SNU PREVENT
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, SeongJoon Koh, Associate Professor, Seoul National University Hospital
Other Study IDs: H-2110-155-1266
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: Crohn Disease; Ulcerative Colitis; Psoriasis; Ankylosing Spondylitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Psoriasis; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to investigate characteristics of individuals at high risk for developing Inflammatory Bowel Disease (IBD) in order to identify risk factors associated with its incidence.

The main question it aims to answer is:

What are the risk factors for developing Inflammatory Bowel Disease?

Researchers will compare groups at high risk for IBD to healthy populations and to patients already diagnosed with IBD.

Participants will

* undergo assessments of general demographic and clinical characteristics.
* be monitored for symptoms using questionnaires administered at regular intervals.
* have blood tests and stool examinations performed. In cases where participants undergo colonoscopy for routine clinical indications, gut biopsies will also be performed.

DETAILED DESCRIPTION:
Recruitment announcements for participants who are first-degree relatives with patients of IBD will be posted on the bulletin board of the patient community, the outpatient bulletin board, and in the consultation room. For patients with confirmed Anti-Saccharomyces cerevisiae antibody (ASCA) positivity or those diagnosed with autoimmune diseases, recruitment will be conducted from among outpatients who meet the criteria. Detailed explanations about the study will be provided, and consent to participate will be obtained prior to recruitment.

Blood and stools will be used for genomic and proteomic, metabolomic analysis. 16s rRNA gene sequencing and whole genome shotgun sequencing will be done for microbiome analysis. Biopsy specimen will be used for proteomic analysis.

Adverse events related with blood sampling will be monitored in outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* first-degree relatives of Inflammatory Bowel Disease patients
* patients who are diagnosed with autoimmune diseases
* patients with functional gastrointestinal disorders who are ASCA-positive

Exclusion Criteria:

* Patients with symptoms such as a 10% weight loss within 3 months, abdominal pain, hematochezia, or diarrhea will undergo colonoscopy, and those diagnosed with Inflammatory Bowel Disease will be excluded.
* Treatment history of Diabetes Mellitus, Irritable Bowel Syndrome, or colon cancer.

Min Age: 10 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals at high risk for Inflammatory Bowel Disease (IBD), including: (1) first-degree relatives of IBD patients who routinely visit the outpatient clinics; (2) individuals with a confirmed positive serum ASCA result identified in the outpatient clinics; and (3) patients with autoimmune diseases who are regularly followed at outpatient clinics. Participants will be recruited from Seoul National University Hospital, Seoul Metropolitan Government-Seoul National University Boramae Medical Center, and Seoul National University Hospital Healthcare System Gangnam Center.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Inflammatory Bowel Disease | Up to 20 years from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea